CLINICAL TRIAL: NCT07007390
Title: Systems Biology of Amyotrophic Lateral Sclerosis (ALS)
Status: Not yet recruiting | Type: Observational
Sponsor: Viome (Industry)
Collaborators: Universidade Federal de Santa Catarina (Other)
Responsible Party: Sponsor
Other Study IDs: V234
Record Dates: First submitted 2025-03-28; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: ALS; ALS (Amyotrophic Lateral Sclerosis)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ALS Cohort: Patients of Dr. Espíndola at UFSC that are diagnosed with ALS and meet the inclusion/exclusion criteria.
- Control Cohort: Those that meet the inclusion/exclusion criteria, do not have ALS, and generally are healthy.

SUMMARY:
The goal of this observational study is to identify molecular features in multiple clinical samples and/or the patient environment that are associated with ALS. Participants will collect biological samples and answer questionnaires regarding their health at each appointment with their ALS practitioner.

ELIGIBILITY:
Inclusion Criteria:

* Patient of Dr. Espíndola at UFSC

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ALS cohort: Patients of Dr. Espíndola at UFSC Control cohort: Participants from the general population
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2030-02-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Molecular features of biological samples that are predictive of ALS progression | We will collect samples and health data from each participant from the time of diagnosis to their death or study termination, whichever comes sooner. Specific time frame: We will collect outcome measures through study completion, an average of 3 years.